CLINICAL TRIAL: NCT01500174
Title: Ultraviolet-C Irradiation in the Management of Pressure Ulcers in People With Spinal Cord Injury: A Randomized, Stratified, Placebo-controlled Trial
Brief Title: Ultraviolet-C Effectiveness in the Management of Pressure Ulcers in People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Ethne L Nussbaum, Principle Investigator, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCI-2007-BDRST-465
Record Dates: First submitted 2011-12-14; First posted 2011-12-28 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Pressure Ulcer
Keywords: skin; decubitus; pressure; sore; spinal cord injury
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active UVC device (Experimental): Three times per week irradiation of wound base and periwound skin
  Interventions: Device: ultraviolet therapy UV254
- Placebo UVC device (Placebo Comparator): Three times per week irradiation of wound base and periwound skin
  Interventions: Device: Placebo ultraviolet therapy UV254

INTERVENTIONS:
Device: ultraviolet therapy UV254 — three times per week until wound closure or patient discharge from hospital
  Arms: active UVC device
Device: Placebo ultraviolet therapy UV254 — Three times per week irradiation of wound base and periwound skin
  Arms: Placebo UVC device

SUMMARY:
The objective of the study is to examine the effectiveness of Ultraviolet-C (UVC) for healing pressure ulcers in people with spinal cord injury. UVC is a form of radiation similar to sunlight but it is normally absorbed in the earth's atmosphere. Participants will be assigned by chance to receive placebo-UVC or real UVC treatment, in addition to receiving wound care according to best practice guidelines. The hypothesis is that UVC-treated wounds will heal at a faster rate than wounds receiving placebo treatment.

Given that pressure ulcers impact on an individual's quality of life, and generate high costs to the overall health care system, further work is needed to explore alternative means of pressure ulcer treatment.

DETAILED DESCRIPTION:
UVC or placebo UVC will be applied to wounds three times per week. Intact skin around the wound edge and the wound base will be irradiated.

ELIGIBILITY:
Inclusion Criteria:

* traumatic, non-traumatic or congenital spinal cord injury C2-L2
* pressure ulcer stage 2 or higher

Exclusion Criteria:

* neoplastic wound
* wound surgically repaired within past 3 months
* wound currently treated with negative pressure therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in ulcer area relative to baseline | At baseline and repeated weekly up to wound closure or duration of hospital stay to a maximum of 32 weeks
  Wounds are photographed at baseline and measurement is repeated every week either until the wound is closed or the subject is discharged from hospital, up to a maximum of 32 weeks. A metric reference is fixed to skin adjacent to the wound. A blinded assessor measures area directly from the number-coded images using digital software. Percent change is calculated each week relative to baseline.

SECONDARY OUTCOMES:
Mean change in ulcer area between consecutive weeks | At baseline and repeated weekly up to wound closure or duration of hospital stay up to a maximum of 32 weeks
  Wounds are photographed at baseline and measurement is repeated every week either until the wound is closed or the subject is discharged from hospital, up to a maximum of 32 weeks. A metric reference is fixed to skin adjacent to the wound. A blinded assessor measures area directly from the number-coded images using digital software. Percent change in area relative to the previous measurement is calculated each week for the individual and then averaged for the individual over all weeks of the study.
Change in Photographic Wound Assessment Tool (PWAT) | From baseline to wound closure or when the subject is discharged from hospital
  The PWAT characterizes six aspects of wound appearance (wound edge, necrotic tissue type and amount, skin colour, granulation tissue and epithelialization), and yields scores ranging from 0-24, where higher scores indicate more severe wounds. A blinded assessor scored the PWAT using the number-coded images.
Change in Cardiff Wound Impact Schedule (CWIS) | From baseline to wound closure or when subject is discharged from hospital
  The CWIS is a condition-specific quality of life (QOL) tool that evaluates wound impact on four domains: overall QOL, well-being, physical experience and the perceived stress of the physical experience.
Follow-up wound status | At 1, 6 and 12 months post-intervention
  Telephone interview - subjects were asked about status of study wounds - open or closed

CONTACTS AND LOCATIONS:
Overall Officials: Ethne L Nussbaum, PhD, Principal Investigator — Toronto Rehabilitation Institute; Colleen F McGillivray, MD, FRCPC, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Nussbaum EL, Biemann I, Mustard B. Comparison of ultrasound/ultraviolet-C and laser for treatment of pressure ulcers in patients with spinal cord injury. Phys Ther. 1994 Sep;74(9):812-23; discussion 824-5. doi: 10.1093/ptj/74.9.812. PMID 8066108
- [Derived] Nussbaum EL, Flett H, Hitzig SL, McGillivray C, Leber D, Morris H, Jing F. Ultraviolet-C irradiation in the management of pressure ulcers in people with spinal cord injury: a randomized, placebo-controlled trial. Arch Phys Med Rehabil. 2013 Apr;94(4):650-9. doi: 10.1016/j.apmr.2012.12.003. Epub 2012 Dec 13. PMID 23246896